CLINICAL TRIAL: NCT06798389
Title: Nurse Follow-up to Reduce Inappropriate Emergency Department Utilization in Adult Patients Seen for Ambulatory Sensitive Conditions in CMSL
Brief Title: CMSL Ambulatory Sensitive Condition Nudge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-1716
Record Dates: First submitted 2025-01-06; First posted 2025-01-29 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Behavioral Intervention; Emergency Department Visits; Nurse Care Coordination
Keywords: Nudge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse Nudge (Experimental): Nurses in CMSL clinics will receive a notification to provide follow-up outreach to patients after the patient receives an ambulatory sensitive diagnosis.
  Interventions: Behavioral: Nurse Nudge
- Control (No Intervention): Nurses in CMSL clinics will receive standard follow-up notifications, which may mean no notifications, after a patient has received an ambulatory sensitive diagnosis.

INTERVENTIONS:
Behavioral: Nurse Nudge — Nurses will be nudged to call the patients, which may increase the likelihood that the patient receives a post-appointment follow-up call.
  Arms: Nurse Nudge

SUMMARY:
The project aims to evaluate a nurse-led intervention to reduce inappropriate emergency department (ED) use among adult patients seen at Geisinger's Community Medicine Service Line (CMSL) clinics. The intervention occurs immediately following an appointment where they received a diagnosis of an ambulatory sensitive condition (ASC). The evaluation will compare eligible patients with an ASC who were randomly assigned to receive follow-up outreach from a nurse (who was automatically prompted via the Epic electronic health record system to initiate outreach) with those who were randomly assigned to receive standard care. Analyses will be intent-to-treat. The primary outcome is ED use in the week following the appointment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years +
* Has a visit in CMSL with an ambulatory sensitive condition (ASC) encounter diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3016 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
ED Visit (yes/no) | within 7 days following day of appointment
  Does outreach decrease ED visits?

OTHER OUTCOMES:
Nurse call to patient | Within 7 days post-appointment
  Does the nurse nudge increase post-appointment nurse calls to patients?

CONTACTS AND LOCATIONS:
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT06798389/Prot_SAP_000.pdf